CLINICAL TRIAL: NCT06766786
Title: Perioperative Magnesium Supplementation in Simultaneous Pancreas-Kidney Transplantation Patients
Brief Title: Magnesium Supplementation in Simultaneous Pancreas-Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Dr Olu Bamgbade, MD, FRCPC (Other)
Collaborators: Central Manchester University Hospitals NHS Foundation Trust (co-sponsor, UK) (Unknown)
Responsible Party: Sponsor-Investigator, Dr Olu Bamgbade, MD, FRCPC, Professor, Salem Anaesthesia Pain Clinic
Organization: Salem Anaesthesia Pain Clinic (Other)
Other Study IDs: SalemAne Magnesia SPK Transpl
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Renal Failure Chronic Requiring Dialysis; Diabetes Mellitus, with Complications; Glomerulosclerosis; Pancreatic Insufficiency (Exocrine and Endocrine); Transplantation, Kidney; Pancreas Transplantation
Keywords: SPK transplant; Simultaneous pancreas-kidney (SPK) transplant; Hypomagnesemia transplantation; Hypomagnesemia kidney transplant; Hypomagnesemia pancreas-kidney transplant; Hypomagnesemia simultaneous pancreas-kidney transplant
MeSH Terms: conditions — Diabetes Complications; Exocrine Pancreatic Insufficiency | interventions — Magnesium Sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic pancreas-kidney failure.: Adult patients with diabetes mellitus and chronic pancreas-kidney failure who require insulin and hemodialysis therapy. Intravenous magnesium supplementation was given intraoperatively to consenting patients receiving simultaneous pancreas-kidney (SPK) transplantation.
  Interventions: Drug: Magnesium Sulfate high dose

INTERVENTIONS:
Drug: Magnesium Sulfate high dose — Patients undergoing simultaneous pancreas-kidney (SPK) transplantation who gave their consent were given an intravenous magnesium supplement at a dose of 45-50 mg/kg over the course of an hour during the procedure.

SUMMARY:
Magnesium is essential in human physiology. Simultaneous pancreas-kidney (SPK) transplant recipients frequently experience hypomagnesemia. The effects of hypomagnesaemia are harmful. This observational study assessed intraoperative magnesium supplementation's utility in patients undergoing SPK transplantation. Perioperative hemodynamics were monitored. Postoperative serum magnesium was monitored at 12 hours and 48 hours.

DETAILED DESCRIPTION:
A vital component of human physiology is magnesium. It is common for recipients of simultaneous pancreas-kidney (SPK) transplants to have hypomagnesemia. The consequences of hypomagnesaemia are detrimental. This prospective observational study evaluated the effectiveness and safety of intraoperative magnesium supplementation in adult SPK transplant recipients. Arrhythmia and perioperative hemodynamics were observed. Serum magnesium levels were checked 12 and 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult diabetic patients who require insulin therapy and hemodialysis due to pancreatic-kidney failure.

Exclusion Criteria:

* Adult diabetic patients who do not require insulin therapy and hemodialysis.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort population of consecutive adult pancreatic-kidney failure patients on regular insulin and hemodialysis therapy and consenting to simultaneous pancreas-kidney (SPK) transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-01-02 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Serum magnesium levels. | 48 hours
  Serum magnesium levels after surgery at 12 and 48 hours.
Perioperative cardiovascular incidents. | 48 hours
  Incidence rate of intraoperative and postoperative dysrhythmia events for each patient.

SECONDARY OUTCOMES:
Postoperative neurological incidents. | 48 hours
  Incidence rate of postoperative confusion, muscle spasms, or weakness in each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Olumuyiwa Bamgbade, MD, FRCPC, Study Director — Salem Anaesthesia Pain Clinic
Locations (1):
- Central Manchester University Hospital, Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared after the research has been analyzed and published.

REFERENCES:
- [Background] Bamgbade OA. Intraoperative magnesium supplementation improves gynecology major surgery perioperative outcome. J Clin Anesth. 2018 Feb;44:21. doi: 10.1016/j.jclinane.2017.10.019. No abstract available. PMID 29100019